CLINICAL TRIAL: NCT05021484
Title: Safety, Tolerability and Efficacy of Monoclonal CD38 Antibody Felzartamab in Late Antibody-Mediated Renal Allograft Rejection - A Phase 2 Pilot Trial
Brief Title: Felzartamab in Late Antibody-Mediated Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Farsad Eskandary (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Alberta (Other); Biogen (Industry)
Responsible Party: Sponsor-Investigator, Farsad Eskandary, Ass. Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EK1161/2021; 2021-000545-40 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-25 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Antibody-mediated Rejection
Keywords: CD38; Kidney transplantation
MeSH Terms: interventions — felzartamab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Felzartamab (Active Comparator): 9 doses of felzartamab as an intravenous infusion over 6 treatment cycles at 28 days each. Dosing occurs every week in cycle 1 and every four weeks in cycles 2-6.
  Interventions: Drug: Felzartamab
- Placebo (Placebo Comparator): 9 doses of placebo as an intravenous infusion over 6 treatment cycles at 28 days each. Dosing occurs every week in cycle 1 and every four weeks in cycles 2-6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Felzartamab — Intravenous infusion in regular intervals over 6 months
  Other Names: MOR202, CD38 monoclonal antibody
  Arms: Felzartamab
Drug: Placebo — Intravenous infusion in regular intervals over 6 months
  Other Names: 0.9% Saline
  Arms: Placebo

SUMMARY:
This prospective trial will assess the safety, tolerability, pharmacokinetics, immunogenicity, pharmacodynamics and efficacy of the fully human CD38 monoclonal antibody felzartamab in kidney transplant recipients with late active or chronic-active ABMR. The study is designed as a randomized, controlled, double-blind pilot phase 2 trial. Participants will be randomized to receive either felzartamab or placebo for a period of six months, and then followed for another six months. After six and twelve months, study participants will be subjected to follow-up allograft biopsies.

DETAILED DESCRIPTION:
This prospective bi-center study (University of Vienna, Charité Universitätsmedizin Berlin; Sponsor: Medical University of Vienna, Vienna, Austria; Funder: MorphoSys AG, Planegg, Germany) is an investigator-driven pilot trial designed to assess the safety&tolerability (primary endpoint), pharmacokinetics, immunogenicity, pharmacodynamics and efficacy (preliminary assessment) of the fully human CD38 monoclonal antibody felzartamab in kidney transplant recipients diagnosed with late active or chronic-active antibody-mediated rejection (ABMR) after kidney transplantation.

Adult renal allograft recipients with anti-HLA donor-specific antibodies (DSA) and biopsy-proven ABMR (Banff 2019 classification) ≥180 days post-transplantation will be identified and recruited at the kidney transplantation outpatient services of the two center sites.

The primary endpoint will be safety and tolerability. Participants will be randomized to receive either felzartamab (intravenous administration) or placebo (1:1 randomization stratified by study site and according to ABMR categories) for a period of 6 months (administration of felzartamab/placebo at day 0, 7, 14, 21, and thereafter in 4-weekly intervals. After six (week 24) and twelve months (week 52), study participants will be subjected to follow-up allograft biopsies.

Primary goals of the trial are to assess the safety, pharmacokinetics and pharmacodynamics (peripheral blood plasma cell and natural killer cell depletion) of a 6-month course of treatment over a period of 12 months. The trial will in addition provide first data on efficacy (progression/activity of rejection, blood biomarkers) and potential associations of treatment with parameters reflecting clinical progression of allograft dysfunction, including the course of estimated glomerular filtration rate.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Age >18 years (maximum: 80 years)
* Functioning living or deceased donor allograft after ≥180 days post-transplantation
* eGFR ≥20 ml/min/1.73 m2 (CKD-EPI formula)
* HLA class I and/or II antigen-specific antibodies (preformed and/or de novo DSA).
* Active or chronic/active ABMR (±C4d in PTC) according to the Banff 2019 classification
* Molecular ABMR score (MMDx) ≥0.2

Exclusion Criteria:

* Patients actively participating in another clinical trial
* Age ≤18 years
* Female subject is pregnant or lactating or not on adequate contraceptive therapy
* ABO-incompatible transplant
* Index biopsy results:
* T-cell-mediated rejection classified Banff grade ≥I
* De novo or recurrent severe thrombotic microangiopathy
* Polyoma virus nephropathy
* De novo or recurrent glomerulonephritis
* Acute rejection treatment ≤3 month before screening
* Previous treatment with other CD38 monoclonal antibodies (e.g. daratumumab)
* Previous treatment with other immunomodulatory monoclonal/polyclonal antibodies (e.g. CD20 Ab rituximab, IL-6/IL-6R Ab) ≤3 months before study treatment
* Total bilirubin >2×the upper limit of normal [ULN], alanine transaminase and aspartate aminotransferase >2·5×ULN
* Haemoglobin <8 g/dL
* Thrombocytopenia: Platelets <100 G/L
* Leukopenia: Leukocytes <3 G/L
* Neutropenia: Neutrophils < 1.5 G/L
* Hypogammaglobulinemia: Serum IgG <400 mg/dL
* Active viral, bacterial or fungal infection precluding intensified immunosuppression
* Active malignant disease precluding intensified immunosuppressive therapy
* Latent or active tuberculosis (positive QuantiFERON-TB-Gold test)
* Administration of a live vaccine within 6 weeks of screening
* History of alcohol or illicit substance abuse
* Serious medical or psychiatric illness likely to interfere with participation in the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 12 months
  (Serious) adverse events will be classified using the Medical Dictionary for Regulatory Activities (MedDRA). Documentation of an AE will include the assessment of its relationship with the study drug (unrelated, related) and the severity of AE will be graded on a three-point scale (mild, moderate, severe).

SECONDARY OUTCOMES:
Felzartamab serum concentration | At day 0, week 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 44, 48 and 52
  Total felzartamab serum concentration (ELISA, ng/mL)
Anti-Felzartamab antibodies | At day 0, week 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 44, 48 and 52
  Concentration of anti-felzartamab antibodies in serum (ELISA, ng/mL)
Morphologic ABMR categories | At week 24 and at week 52
  Phenotyping of renal transplant biopsies: active ABMR vs. chronic active ABMR vs. chronic inactive ABMR
Serum donor-specific antibody (DSA) levels | Week 0, 12, 24, and 52
  Mean fluorescence intensity (MFI) of the immunodominant DSA (Luminex)
Serum immunoglobulin levels | Week 0, 12, 24, and 52
  Ig (sub)classes (ELISA, Nephelometry, mg/dL)
Leukocyte subsets in peripheral blood | Week 0, 1, 4, 8, 12, 24, and 52
  Counts of circulating plasma cells, natural killer cells, T and B cell subpopulations (flow cytometry, cell counts)
Immunologic biomarkers | Week 0, 12, 24, and 52
  CXCL9 and CXCL10 levels in blood and urine, BAFF levels in blood (ELISA, Luminex)
Torque Teno virus | Week 0, 12, 24, and 52
  Torque Teno virus (TTV) levels in plasma (quantitative PCR)
eGFR | At day 0, week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 44, 48 and 52
  Estimated GFR (CKD-EPI, mL/min/1.73m2)
Proteinuria | At day 0, week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 44, 48 and 52
  Urinary protein excretion in spot urine (protein/creatinine ratio in mg/g)
Graft loss | 12 months
  Graft failure: time (months) to event (Kaplan Meier)
Death | 12 months
  Patient death: time (months) to event (Kaplan Meier)
Glomerulitis plus peritubular capillaritis sum score | At week 24 and at week 52
  Grading of renal transplant biopsies using a semiquantitative score (g+ptc 0-6); higher = worse prognosis
Transplant glomerulopathy score | At week 24 and at week 52
  Grading of renal transplant biopsies using a semiquantitative score (cg 0-3); higher = worse prognosis
C4d score | At week 24 and at week 52
  Grading of renal transplant biopsies using a semiquantitative score (c4d 0-3); higher = worse prognosis
Molecular ABMR score | At week 24 and at week 52
  ABMR score (0.0-1.0, dimensionless number) assessed via the Molecular Microscope Diagnostic Platform (MMDx); higher = worse prognosis
Molecular ABMR categories | At week 24 and at week 52
  Molecular archetype analysis of rejection phenotypes using the Molecular Microscope Diagnostic Platform (MMDx). Phenotypes: early-stage ABMR; fully developed ABMR; late-stage ABMR

CONTACTS AND LOCATIONS:
Overall Officials: Georg A Böhmig, MD, Principal Investigator — Department of Internal Medicine III, Medical University of Vienna
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Charité University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doberer K, Klager J, Gualdoni GA, Mayer KA, Eskandary F, Farkash EA, Agis H, Reiter T, Reindl-Schwaighofer R, Wahrmann M, Cohen G, Haslacher H, Bond G, Simonitsch-Klupp I, Halloran PF, Bohmig GA. CD38 Antibody Daratumumab for the Treatment of Chronic Active Antibody-mediated Kidney Allograft Rejection. Transplantation. 2021 Feb 1;105(2):451-457. doi: 10.1097/TP.0000000000003247. PMID 32235256
- [Background] Raab MS, Engelhardt M, Blank A, Goldschmidt H, Agis H, Blau IW, Einsele H, Ferstl B, Schub N, Rollig C, Weisel K, Winderlich M, Griese J, Hartle S, Weirather J, Jarutat T, Peschel C, Chatterjee M. MOR202, a novel anti-CD38 monoclonal antibody, in patients with relapsed or refractory multiple myeloma: a first-in-human, multicentre, phase 1-2a trial. Lancet Haematol. 2020 May;7(5):e381-e394. doi: 10.1016/S2352-3026(19)30249-2. Epub 2020 Mar 11. PMID 32171061
- [Background] Mayer KA, Doberer K, Eskandary F, Halloran PF, Bohmig GA. New concepts in chronic antibody-mediated kidney allograft rejection: prevention and treatment. Curr Opin Organ Transplant. 2021 Feb 1;26(1):97-105. doi: 10.1097/MOT.0000000000000832. PMID 33315763
- [Derived] Madill-Thomsen KS, Gauthier PT, Abouljoud M, Bhati C, Bruno D, Ciszek M, Durlik M, Feng S, Foroncewicz B, Grat M, Jurczyk K, Levitsky J, McCaughan G, Maluf D, Montano-Loza A, Moonka D, Mucha K, Myslak M, Perkowska-Ptasinska A, Piecha G, Reichman T, Tronina O, Wawrzynowicz-Syczewska M, Zeair S, Halloran PF. Defining an NK Cell-enriched Rejection-like Phenotype in Liver Transplant Biopsies From the INTERLIVER Study. Transplantation. 2025 Aug 1;109(8):1367-1382. doi: 10.1097/TP.0000000000005269. Epub 2025 Jan 9. PMID 39780312
- [Derived] Mayer KA, Schrezenmeier E, Diebold M, Halloran PF, Schatzl M, Schranz S, Haindl S, Kasbohm S, Kainz A, Eskandary F, Doberer K, Patel UD, Dudani JS, Regele H, Kozakowski N, Klager J, Boxhammer R, Amann K, Puchhammer-Stockl E, Vietzen H, Beck J, Schutz E, Akifova A, Firbas C, Gilbert HN, Osmanodja B, Halleck F, Jilma B, Budde K, Bohmig GA. A Randomized Phase 2 Trial of Felzartamab in Antibody-Mediated Rejection. N Engl J Med. 2024 Jul 11;391(2):122-132. doi: 10.1056/NEJMoa2400763. Epub 2024 May 25. PMID 38804514
- [Derived] Mayer KA, Budde K, Halloran PF, Doberer K, Rostaing L, Eskandary F, Christamentl A, Wahrmann M, Regele H, Schranz S, Ely S, Firbas C, Schorgenhofer C, Kainz A, Loupy A, Hartle S, Boxhammer R, Jilma B, Bohmig GA. Safety, tolerability, and efficacy of monoclonal CD38 antibody felzartamab in late antibody-mediated renal allograft rejection: study protocol for a phase 2 trial. Trials. 2022 Apr 8;23(1):270. doi: 10.1186/s13063-022-06198-9. PMID 35395951